CLINICAL TRIAL: NCT01675323
Title: Glutamate, Hyperarousal and Restless Legs Syndrome
Status: Completed | Type: Observational
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Richard Allen, Research Associate, Department of Neurology, Johns Hopkins University
Other Study IDs: NA_00073951
Record Dates: First submitted 2012-08-27; First posted 2012-08-29 (Estimated); Last update posted 2017-03-01 (Actual); Status verified 2017-02

CONDITIONS: Restless Legs Syndrome
Keywords: Restless Legs Syndrome; RLS
MeSH Terms: conditions — Restless Legs Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood and urine (female participants only)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- RLS Patients: Participants who have diagnosed RLS with diagnosis confirmed by study investigators.
- Healthy Controls: Participants without RLS who are generally healthy and matched for gender, age, educational level, and race to patients in the RLS group.

SUMMARY:
Restless Legs Syndrome (RLS) research has focused on the sensory features and failed to address an important aspect of RLS; i.e. a 'hyperarousal' or profound chronic sleep loss without significant excessive daytime sleepiness. This hyperarousal produces RLS symptoms by overwhelming the normal inhibitory processes needed to decrease sensory and motor cortical activity for resting and sleep. Thus the hyperarousal produces both the RLS need to move when trying to rest and the inability to maintain sleep. The biological consequences of this hyperarousal process on sleep (increased wake time) and cortical excitability (as demonstrated by transcranial magnetic stimulation (TMS)) are postulated to reflect increased degree of excitatory glutamatergic activity, and therefore affected brain regions will show relatively increased glutamate (Glu) and glutamine (Gln) on MR spectroscopy (MRS). Changes in inhibitory activity and GABA may also occur, but less significantly than the increase in Glu/Gln. Our pilot MRS data discovered a new abnormality in RLS: increased Thalamic Glx (Glu + Gln) that correlated well with sleep measures of hyperarousal. Glx levels are not specific for the neurotransmitter role of Glu.

In this project RLS and matching controls subjects will be studied using polysomnograms (PSG) and TMS and 7T MRI for MRS that provides accurate measurement of Gln levels, which reflect mostly neurotransmitter Glu activity. The first aim is to confirm that Gln is increased in the thalamus and to determine if this also occurs in the motor and sensory cortices. The relation between Glu, Gln and GABA will also be evaluated. Second, assessments will be made of the degree of relation between Gln increase and the hyperarousal effects on sleep and cortical excitability (TMS). This would demonstrate that abnormally increased Glu activity is primary to RLS hyperarousal and radically changes the emphasis in RLS to be less on dopamine and more on Glu-hyperarousal as a major feature of RLS.This is an entirely new direction for RLS research and treatment development. The new concept of hyperarousal adds a missing dimension to understanding RLS, namely the discovery of the Glu abnormality and its central relation to the other hyperarousal features.

DETAILED DESCRIPTION:
Moderate to severe Restless Legs Syndrome (RLS) is a major public health problem, significantly affecting 1.5 to 3% of adult Americans (3 - 7 million), resulting in profound sleep loss and an urge to move during sitting or resting in the later part of the day. Work productivity is decreased by 20%, quality of life is as bad or worse than that for other chronic diseases, e.g. arthritis and diabetes, and there is increased cardio-vascular disease risk. Current approved dopaminergic treatments fail to improve sleep time, engender impulsive behaviors and may make RLS worse. New treatments and new research directions to find them are needed. The current research focus on the sensory features has failed to address an important aspect of RLS; i.e. a 'hyperarousal' or profound chronic sleep loss without significant excessive daytime sleepiness. This hyperarousal produces RLS symptoms by overwhelming the normal inhibitory processes needed to decrease sensory and motor cortical activity for resting and sleep. Thus the hyperarousal produces both the RLS need to move when trying to rest and the inability to maintain sleep. The biological consequences of this hyperarousal process on sleep (increased wake time) and cortical excitability (as demonstrated by transcranial magnetic stimulation (TMS)) are postulated to reflect increased degree of excitatory glutamatergic activity, and therefore affected brain regions will show relatively increased glutamate (Glu) and glutamine (Gln) on MR spectroscopy (MRS). Changes in inhibitory activity and GABA may also occur, but less significantly than the increase in Glu/Gln. Our pilot MRS data discovered a new abnormality in RLS: increased Thalamic Glx (Glu + Gln) that correlated well with sleep measures of hyperarousal. Glx levels are not specific for the neurotransmitter role of Glu. In this project RLS and matching controls subjects will be studied using polysomnograms (PSG) and TMS and 7T MRI for MRS that provides accurate measurement of Gln levels, which reflect mostly neurotransmitter Glu activity. The first aim is to confirm that Gln is increased in the thalamus and to determine if this also occurs in the motor and sensory cortices. The relation between Glu, Gln and GABA will also be evaluated. Second, assessments will be made of the degree of relation between Gln increase and the hyperarousal effects on sleep and cortical excitability (TMS). This would demonstrate that abnormally increased Glu activity is primary to RLS hyperarousal and radically changes the emphasis in RLS to be less on dopamine and more on Glu-hyperarousal as a major feature of RLS. This is an entirely new direction for RLS research and treatment development. The new concept of hyperarousal adds a missing dimension to understanding RLS, namely the discovery of the Glu abnormality and its central relation to the other hyperarousal features. It opens the opportunity to develop new animal and cell RLS research. It provides new directions for medication treatment development, changes the emphasis for primary treatment toward Glu drugs and the MRS provides a useful and accessible measure for evaluating medication treatment benefits.

ELIGIBILITY:
Inclusion Criteria:

* All subjects

  1. 18 years or older
  2. Normal mental status and able to give informed consent.
  3. Regular sleep times start between 21:00 and 01:00 5 out of 7 days a week
  4. General good health and ambulatory
* RLS patients

  1. Diagnosis of primary RLS confirmed by the PI or Dr. Earley
  2. History indicating if RLS symptoms were not treated, thy would for the last 6 months

     1. Occur at least 5 out of 7 days a week
     2. Almost always disrupt sleep
  3. For phase 2 admission to the Clinical Research Unit: Home screening on a clinical log shows RLS symptoms for at least 5 of 7 days, IRLS score at the end of home monitoring ≥ 15 and PAM-RL measures show average PLMS/hr ≥15.
* Control subjects

  1. No history of any of the 4 essential criteria for diagnosis of RLS (1).
  2. For phase 2 admission to the Clinical Research Unit: Home screening on the PAM-RL indicates average PLMS/hr ≤ 10 and the sleep-wake log shows regular times in bed between 21:00 and 01:00 bed times with 6.0 to 10.0 hours in bed for 5 out of for 7 nights.

Exclusion Criteria:

* All subjects

  1. Major mental history as determined by history
  2. Clinically significant sleep apnea on prior PSG or on screening first night PSG (apnea/hypopnea rate >15/hr).
  3. Any medical or neurological disorder other than RLS likely to compromise normal sleep, interfere with interpretation of results, or would place the subject at risk when participating in the study (e.g. Chronic pain, dementia, ALS, stroke, MS, untreated thyroid).
  4. Any use of DA antagonists for more than one week in the past 6 months, other than for nausea.
  5. Women who are pregnant or lactating or at risk for getting pregnant (not using appropriate birth control nor post-menopausal).
  6. Failure to have clear hand dominance, ambidextrous as assessed by the Edinburgh Handedness Inventory (Could influence outcomes on TMS).
  7. Musicians and professional typists (Might influence performance on TMS measure)
  8. A significant neurological disorder (such as stroke, Parkinson's Disorder, Multiple Sclerosis) that could impair fine motor performance.
  9. Metal in the body (e.g., pacemakers, implantable pumps, stimulators, orthodontics, etc) that would cause problems for the MRI or TMS.
  10. Medication use that would alter sleep including any GABA active medications and any anti- depressants or other significant psychiatric medications or medications that would affect Glu.
  11. History of claustrophobia or problems with closed MRI scans not resolved.
  12. History of vertigo, seizure disorder, middle-ear disorder, or double vision.
  13. Body size not compatible with using T7 MRI.
* RLS patients

  1. History of clinically significant sleep disorder other than that with RLS.
  2. Medical disorder or current medication use that exacerbates or might have started the RLS
* Control subjects

  1. History of clinically significant sleep disorder including insomnia (primary or psycho-physiological)
  2. Score on the Pittsburgh Sleep Quality Inventory (PSQI) >5
  3. Family history indicating possible RLS in a first-degree relative

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects with RLS and healthy subjects, 18 years of age or older, matched for age, gender, race, and educational level. Both men and women will be included.
Sampling Method: Non-Probability Sample
Enrollment: 77 (Actual)
Dates: Start 2012-08; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
MR Spectroscopy - Glutamate | 2nd Day of Phase 2
  Study of thalamic glutamate levels in the brain using MR Spectroscopy
MR Spectroscopy - GABA | 2nd Day of Phase 2
  Study of thalamic GABA levels in the brain using MR Spectroscopy

CONTACTS AND LOCATIONS:
Overall Officials: Richard Allen, Ph.D., Principal Investigator — Johns Hopkins University
Locations (2):
- United States (2):
  - Johns Hopkins Baview Medical, Baltimore, Maryland
  - Johns Hopkins Bayview Medical Campus, Baltimore, Maryland